CLINICAL TRIAL: NCT04784897
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Brilacidin in Hospitalized Participants With COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of Brilacidin in Hospitalized Participants With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovation Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI-BRIc-201
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; coronavirus; Brilacidin; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — brilacidin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brilacidin + SoC (Experimental): Brilacidin IV infusion, 3 days and up to 5 days, in addition to Standard of Care
  Interventions: Drug: Brilacidin; Drug: Standard of Care (SoC)
- Placebo + SoC (Placebo Comparator): Placebo IV infusion, 3 days and up to 5 days, in addition to Standard of Care
  Interventions: Drug: Placebo; Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: Brilacidin — Brilacidin IV infusion
  Arms: Brilacidin + SoC
Drug: Placebo — Placebo IV infusion
  Arms: Placebo + SoC
Drug: Standard of Care (SoC) — SoC therapies for COVID-19

SUMMARY:
The study assessed the efficacy and safety of Brilacidin for the treatment of COVID-19 in hospitalized participants

DETAILED DESCRIPTION:
This Phase 2 study was a randomized, blinded, placebo-controlled, parallel group design.

The target population treated were patients with moderate to severe COVID-19, active SARS-CoV-2 infection confirmed by positive standard polymerase chain reaction (PCR) test (or equivalent/ other approved diagnostic test) within 4 days prior to starting study treatment, and were hospitalized with respiratory distress but not yet requiring high-level respiratory support (as defined in exclusion criterion #2). See inclusion/exclusion criteria.

For each participant, the study was comprised of three parts:

1. Screening/ Baseline visit (Day -1 to 1): Lasting up to 24-48 hours and comprised screening/ baseline assessments. This visit was to confirm that study inclusion and exclusion criteria were met by participants prior to randomization.
2. Treatment period (Day 1-3 or Day 1-5): Randomized subjects received blinded study treatment once daily for 3 or 5 days by IV infusion, in addition to Standard of Care (SoC).
3. Follow-up period (Day 4 or 6 through Day 60): Subjects were assessed daily while hospitalized. Discharged patients were asked to attend study visits at Days 15 and 29. A follow-up visit at Day 60(±10), by telephone call, was performed to confirm patient status.

All participants had a series of efficacy and safety assessments performed, including laboratory assays. Additional blood samples and nasopharyngeal (NP) swabs were also obtained (oropharyngeal (OP) swabs were to be collected only in exceptional circumstances).

Study participants/subjects were randomized to active or placebo, and the study started with 3 days of study drug administration. After an interim analysis safety review, by an independent Data Monitoring Committee (DMC), dosing was extended to 5 days. Hence, subjects recruited after the interim analysis received 5 days of study treatment.

For study analyses, subjects randomized to placebo were pooled since duration of placebo should not impact efficacy or safety outcomes. As the different treatment durations for Brilacidin have potential to impact efficacy and/or safety outcomes, 3-dose and 5-dose active arms were analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written Informed Consent Form (ICF) to participate in the clinical study by patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representative.
* Male or non-pregnant female adults between 18 and 80 years of age, inclusive, at time of informed consent.
* SARS-CoV-2 infection confirmed by positive standard polymerase chain reaction (PCR) test (or equivalent/ other approved diagnostic test) ≤ 4 days before randomization.
* Currently hospitalized and requiring medical care for COVID-19.
* Moderate OR severe COVID-19, defined by respiratory function at screening, as below:

  * Moderate, meets at least one of the following criteria:

    * Peripheral oxygen saturation SpO2 > 93% on room air;
    * Respiratory rate ≥ 20 to < 30 breaths per minute.
  * Severe, meets at least one of the following criteria:

    * Peripheral oxygen saturation SpO2 ≤ 93% on room air OR arterial oxygen partial pressure (PaO2) / fraction of inspired oxygen (FiO2) < 300mmHg (1mmHg=0.133kPa) [corrective formulation should be used for higher altitude regions (over 1000m)];
    * Respiratory rate ≥ 30 breaths per minute.
* Body mass index (BMI) of ≥18 to <40kg/m2 at screening.
* Agrees to the collection of nasopharyngeal (NP) swabs and venous blood per protocol.
* In the opinion of the investigator, willing and able to comply with the study protocol assessments, and is committed to the study and the study follow up visits.

Exclusion Criteria:

* Participation in any other clinical trial of an experimental agent treatment.
* Requiring invasive mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO) at the time of randomization.
* Has explicitly expressed the wish not to receive intensive care support (Do not resuscitate or Do not intubate order) should this become necessary.
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 72 hours, irrespective of the provision of treatment, such as rapidly progressive multiorgan failure.
* Requiring systemic anti-infective therapy for suspected or confirmed active bacterial/fungal/viral systemic infection other than COVID-19.
* Hypertensive urgency (e.g., SBP >220 mmHg or DBP >120 mmHg) or hypertensive emergency within the last 72 hours, as assessed by the investigator following local guidelines.
* If has a history of hypertension in the last 3 months, must have been receiving appropriate anti-hypertensive therapy in accordance with local guidelines.
* Evidence of moderate or severe hepatic impairment (Child-Pugh Class B or C).
* Estimated GFR (eGFR) <30 mL/min/1.73m2 (based on CKD-EPI formula).
* Prior to a participant's study entry, known allergies or intolerance to Brilacidin or formulation excipients.
* Any serious medical or psychiatric condition or test abnormality(ies) that, in the investigator's judgment, puts the participant at significant risk, could confound the study results, or may interfere significantly with the subject's safe participation in and completion of the study.
* Pregnancy or breast-feeding, or positive urine or serum pregnancy test in a pre-dose assessment.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception throughout the study and for up to 30 days after stopping treatment.
* Sexually active males with female partners of childbearing potential unwilling to use a condom when engaging in intercourse of reproductive potential throughout the study and for up to 30 days after stopping treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Innovation Pharmaceuticals Inc., Study Director — Innovation Pharmaceuticals, Inc.
Locations (7):
- United States (2):
  - IPI Investigator Site, Winfield, Illinois
  - IPI Investigator Site, Toledo, Ohio
- Russia (5):
  - IPI Investigator Site, Barnaul
  - IPI Investigator Site, Moscow
  - IPI Investigator Site, Nizniy Novgorod
  - IPI Investigator Site, Pushkin
  - IPI Investigator Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study participants were randomized to active or placebo, and dependent upon if prior to or after the scheduled interim safety analysis, were randomized to 3 days or 5 days of study treatment.
  For study analyses, subjects randomized to placebo were pooled since duration of placebo should not impact efficacy or safety outcomes. As the different treatment durations for Brilacidin have potential to impact efficacy and/or safety outcomes, 3-dose and 5-dose active arms were analyzed separately.
Groups:
- Pooled Placebo + SoC: Saline IV infusion, 3 to 5 daily doses, in addition to Standard of Care..
- Brilacidin 3-dose + SoC: Brilacidin IV infusion, 3 daily doses, in addition to Standard of Care.
- Brilacidin 5-dose + SoC: Brilacidin IV infusion, 5 daily doses, in addition to Standard of Care.
Period: Overall Study
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Started | 60 | 16 | 44
Completed | 56 | 14 | 42
Not Completed | 4 | 2 | 2
Not completed — Death | 4 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study participants were randomized to active or placebo, and dependent upon if prior to or after the scheduled interim safety analysis, were randomized to 3 days or 5 days of study treatment.
  Subjects randomized to placebo are pooled for the analyses since duration of placebo should not impact efficacy or safety outcomes. As the different treatment durations for Brilacidin have potential to impact efficacy and/or safety outcomes, 3-dose and 5-dose active arms were analyzed separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC | Total
Number analyzed (Participants) | 60 | 16 | 44 | 120
Age, Continuous [Mean (Full Range); unit: years] | 58.1 [23 to 77] | 61.4 [44 to 77] | 56.2 [23 to 80] | 57.8 [23 to 80]
Age, Customized [Count of Participants; unit: Participants]
  <=65 years | 40 | 10 | 30 | 80
  >65 years | 20 | 6 | 14 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 8 | 16 | 55
  Male | 29 | 8 | 28 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 59 | 15 | 44 | 118
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 59 | 16 | 43 | 118
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 0 | 3
  Russia | 59 | 14 | 44 | 117
COVID-19 Severity [Count of Participants; unit: Participants]
  Moderate | 24 | 6 | 16 | 46
  Severe | 36 | 10 | 28 | 74
Breathing Status [Count of Participants; unit: Participants]
  Room Air | 21 | 7 | 14 | 42
  Low Flow O2 | 36 | 7 | 29 | 72
  High Flow O2 | 2 | 1 | 1 | 4
  CPAP/BiPAP | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Recovery Through Day 29
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the clinical status ordinal scale with response sustained through Day 29:
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than for per protocol dosing or assessments, as appropriate); 7. Not hospitalized, limitation on activities and/or requiring home oxygen; 8. Not hospitalized, no limitations on activities
Time Frame: Day 1 through Day 29
Population: Intent-to-Treat (ITT) population, which includes all subjects who were randomized and receive at least one dose of study drug; subjects analyzed according to the treatment group to which they were randomized.
  For analyses, placebo subjects were pooled whereas the 3-dose and 5-dose active arms were analyzed separately.
  Censoring: Subjects not achieving recovery, lost to follow-up (for this endpoint) prior to achieving recovery, or who died prior to Day 29, were censored at Day 29.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
days | 12.00 [9.00 to 14.00] | 13.00 [9.00 to 16.00] | 13.00 [11.00 to 14.00]
Statistical Analysis 1: Comparison: Pooled Placebo + SoC vs Brilacidin 5-dose + SoC; Main comparison is between Brilacidin 5-dose and Pooled Placebo; Test type: Superiority; p = 0.7273, Log Rank; Cox Proportional Hazard = 0.9289, 90% CI 2-sided [0.6585 to 1.3102]
Statistical Analysis 2: Comparison: Pooled Placebo + SoC vs Brilacidin 3-dose + SoC; Secondary comparison between Brilacidin 3-dose and Pooled Placebo; Test type: Superiority; p = 0.5975, Log Rank; Cox Proportional Hazard = 0.8968, 90% CI 2-sided [0.5464 to 1.4720]

2. Primary Outcome: Percentage of Participants With Sustained Recovery Through Day 29
Description: as for outcome 1
Time Frame: Day 5, Day 8, Day 11, Day 15, Day 29
Population: ITT population. For analyses, placebo subjects were pooled whereas the 3-dose and 5-dose active arms were analyzed separately.
  Censoring: Subjects not achieving recovery, lost to follow-up (for this endpoint) prior to achieving recovery, or who died prior to Day 29, were censored at Day 29.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
percentage of participants
  By Day 5 | 8.33 | 6.25 | 4.55
  By Day 8 | 25.00 | 18.75 | 20.45
  By Day 11 | 43.33 | 31.25 | 34.09
  By Day 15 | 65.00 | 62.50 | 65.91
  By Day 29 | 90.00 | 87.50 | 93.18

3. Secondary Outcome: Number and Percentage of Participants Achieving Recovery Status Scores at Day 29
Description: Recovery status scores are the following three categories from the clinical status ordinal scale:
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than for per protocol dosing or assessments, as appropriate); 7. Not hospitalized, limitation on activities and/or requiring home oxygen; 8. Not hospitalized, no limitations on activities
Time Frame: Day 29
Population: ITT population. For analyses, placebo subjects were pooled whereas the 3-dose and 5-dose active arms were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants | 54 | 14 | 41

4. Secondary Outcome: Number and Percentage of Participants Who Die or Develop Respiratory Failure by Day 29
Description: Composite endpoint, defined as: Death OR Respiratory failure (requires invasive mechanical ventilation)
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants | 3 | 2 | 2

5. Secondary Outcome: Subject Clinical Status
Description: Clinical status was measured with an 8-point ordinal scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low-flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than for per protocol dosing or assessments, as appropriate)
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 1, Day 8, Day 15, Day 29
Population: ITT population. No. of participants at each timepoint is the sum across all 8 categories of the scale.
  For analyses, placebo subjects were pooled whereas the 3-dose and 5-dose active arms were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants
  Baseline (Day 1): Score 1 | 0 | 0 | 0
  Baseline (Day 1): Score 2 | 0 | 0 | 0
  Baseline (Day 1): Score 3 | 4 | 2 | 1
  Baseline (Day 1): Score 4 | 35 | 7 | 29
  Baseline (Day 1): Score 5 | 21 | 7 | 14
  Baseline (Day 1): Score 6 | 0 | 0 | 0
  Baseline (Day 1): Score 7 | 0 | 0 | 0
  Baseline (Day 1): Score 8 | 0 | 0 | 0
  Day 8: Score 1 | 1 | 0 | 0
  Day 8: Score 2 | 0 | 1 | 0
  Day 8: Score 3 | 4 | 2 | 2
  Day 8: Score 4 | 15 | 1 | 12
  Day 8: Score 5 | 23 | 9 | 20
  Day 8: Score 6 | 2 | 1 | 1
  Day 8: Score 7 | 3 | 1 | 3
  Day 8: Score 8 | 12 | 1 | 6
  Day 15: Score 1 | 1 | 1 | 1
  Day 15: Score 2 | 1 | 0 | 0
  Day 15: Score 3 | 3 | 1 | 1
  Day 15: Score 4 | 5 | 1 | 5
  Day 15: Score 5 | 11 | 3 | 8
  Day 15: Score 6 | 0 | 1 | 5
  Day 15: Score 7 | 4 | 1 | 3
  Day 15: Score 8 | 35 | 8 | 21
  Day 29: Score 1 | 3 | 2 | 2
  Day 29: Score 2 | 0 | 0 | 0
  Day 29: Score 3 | 2 | 0 | 0
  Day 29: Score 4 | 1 | 0 | 1
  Day 29: Score 5 | 0 | 0 | 0
  Day 29: Score 6 | 0 | 0 | 0
  Day 29: Score 7 | 2 | 1 | 1
  Day 29: Score 8 | 52 | 13 | 40

6. Secondary Outcome: Number and Percentage of Participants Achieving at Least One Category Improvement in Clinical Status
Description: as for outcome 5
Time Frame: Day 8, Day 15, Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants
  Day 8 | 30 | 6 | 20
  Day 15 | 44 | 12 | 35
  Day 29 | 55 | 14 | 41

7. Secondary Outcome: Number and Percentage of Participants Achieving at Least Two Category Improvement in Clinical Status
Description: as for outcome 5
Time Frame: Day 8, Day 15, Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants
  Day 8 | 16 | 3 | 10
  Day 15 | 39 | 9 | 27
  Day 29 | 54 | 14 | 41

8. Secondary Outcome: Time to at Least One Category Improvement in Clinical Status
Description: Day to achieving improvement of one or more category on 8-point clinical status ordinal scale.
  Clinical status scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low-flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than for per protocol dosing or assessments, as appropriate)
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
days | 7.00 [6.00 to 9.00] | 10.00 [5.00 to 13.00] | 8.00 [6.00 to 11.00]

9. Secondary Outcome: Time to at Least Two Category Improvement in Clinical Status
Description: Day to achieving improvement of two or more categories on 8-point clinical status ordinal scale.
  Clinical status scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low-flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than for per protocol dosing or assessments, as appropriate)
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
days | 12.50 [9.00 to 14.00] | 14.00 [10.00 to 17.00] | 13.00 [11.00 to 14.00]

10. Secondary Outcome: Time to a National Early Warning Score 2 (NEWS2) of <= 2 Maintained for 24 Hours
Description: Time (in days) from randomization to achieve a NEWS2 score lower or equal to 2 being maintained for at least one 24-hour period.
  NEWS2 was assessed twice daily while hospitalized; if one of the components of the NEWS2 was missing at a particular time point, the NEWS2 was not calculated.
  The National Early Warning Score 2 (NEWS2) assesses a participant's degree of illness as assessed by clinical risk prediction categories based on a set of 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0 to 3 was allocated to each parameter except supplemental oxygen use (score of 0 [no] or 2 [yes]) and level of consciousness (score of 0 [alert, normal health condition] or 3 [altered mental state/confusion, worst health condition]). All parameter scores were summed to get an aggregate NEWS2. NEWS2 ranges from 0 to 20, with higher scores meaning more severity/higher clinical risk
Time Frame: Day 1 through Day 29
Population: ITT population. For analyses, placebo subjects were pooled whereas the 3-dose and 5-dose active arms were analyzed separately.
  NEWS2 Censoring: Subjects with baseline score of 3 or higher, who did not reach NEWS2 of <=2 by Day 29, were censored at last available assessment. Subjects who died were censored on date of death. For those subjects with a baseline score of <=2, subjects were censored at baseline.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 30 | 8 | 26
days | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 5.00]

11. Secondary Outcome: Percentage of Participants Achieving a National Early Warning Score 2 (NEWS2) of <= 2 Maintained for 24 Hours
Description: The National Early Warning Score 2 (NEWS2) assesses a participant's degree of illness as assessed by clinical risk prediction categories based on a set of seven (7) clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0 to 3 was allocated to each parameter except supplemental oxygen use (score of 0 [no] or 2 [yes]) and level of consciousness (score of 0 [alert, normal health condition] or 3 [altered mental state/confusion, worst health condition]). All parameter scores were summed to get an aggregate NEWS2 assessment. Scoring for NEWS2 ranges from 0 to 20, with higher scores meaning more severity/higher clinical risk: low risk (score 1 to 4); low to medium risk (score of 3 in any individual parameter); medium risk (score 5 to 6); high risk (score 7 to 20).
Time Frame: Day 5, Day 8, Day 11, Day 15
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 30 | 8 | 26
percentage of participants
  By Day 5 | 65.62 | 72.73 | 62.07
  By Day 8 | 78.12 | 72.73 | 84.83
  By Day 11 | 84.37 | 72.73 | 94.94
  By Day 15 | 87.50 | 72.73 | 94.94

12. Secondary Outcome: Change From Baseline in National Early Warning Score 2 (NEWS2)
Description: as for outcome 11
Time Frame: Day 1 through Day 29
Population: as for outcome 10
Measure: Mean (Standard Error); unit: score
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
score
  Day 3 | -0.433 (0.225) | -1.000 (0.524) | -0.682 (0.200)
  Day 5 | -1.150 (0.224) | -1.500 (0.769) | -1.455 (0.301)
  Day 8: number analyzed (Participants) | 53 | 15 | 39
  Day 8 | -1.302 (0.262) | -1.400 (0.804) | -1.923 (0.341)
  Day 11: number analyzed (Participants) | 36 | 12 | 30
  Day 11 | -1.472 (0.305) | -2.167 (0.824) | -2.400 (0.436)
  Day 15: number analyzed (Participants) | 58 | 15 | 42
  Day 15 | -1.931 (0.285) | -2.133 (0.940) | -2.619 (0.330)
  Day 29: number analyzed (Participants) | 56 | 12 | 41
  Day 29 | -2.339 (0.243) | -2.667 (0.620) | -3.073 (0.311)

13. Secondary Outcome: Number and Percentage of Participants With Treatment-Emergent Adverse Events
Description: Treatment-Emergent Adverse Events (TEAEs) have onset dates on or after the study treatment start date
Time Frame: Day 1 through Day 60
Population: Safety population, which includes all subjects in the ITT population; subjects in this population analyzed according to treatment received.
  Subjects treated with placebo were pooled for analyses since duration of placebo should not impact outcomes. As the different treatment durations for Brilacidin have potential to impact outcomes, 3-dose and 5-dose active arms were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants
  At least one TEAE | 39 | 14 | 39
  At least one Grade 3 (Severe) TEAE | 9 | 6 | 7
  At least one Grade 4 (Life-threatening) TEAE | 3 | 2 | 0
  At least one Grade 5 (Fatal) TEAE | 4 | 2 | 2

14. Secondary Outcome: Number and Percentage of Participants With Treatment-Emergent Adverse Events of Special Interest
Description: Treatment-Emergent adverse events have onset dates on or after the study treatment start date.
  Adverse Events of Special Interest (AESIs) are (i) hypertension Grade 3 or greater, and (ii) paresthesias / dysesthesias Grade 2 or greater, in accordance with CTCAE (version 5.0) criteria.
Time Frame: Day 1 through Day 60
Population: Safety population. Subjects treated with placebo were pooled for analyses since duration of placebo should not impact outcomes. As the different treatment durations for Brilacidin have potential to impact outcomes, 3-dose and 5-dose active arms were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants
  At least one TEAE of special interest: hypertension Grade 3 or greater | 2 | 3 | 2
  At least one TEAE of special interest: paresthesias/dysesthesias Grade 2 or greater | 0 | 3 | 4

15. Other Pre Specified Outcome: 28-Day Mortality Rate
Description: Incidence of death during the 28 days after start of study treatment
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 60 | 16 | 44
Participants | 3 | 2 | 2

16. Post Hoc Outcome: Time to Sustained Recovery Through Day 29 for Participant Sub-group With C-Reactive Protein (CRP) in the Highest Quartile (4th Quartile) at Baseline
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: Pooled Placebo vs Brilacidin 5-dose arm analyzed, for Post-hoc Per Protocol (PP) CRP sub-group.
  Post-hoc PP population is a subset of ITT population with the following differences:
  * Excludes subjects with viral load <10 copies/mL (i.e., below lower limit of quantitation) at baseline
  * Excludes subjects with <3 days of study drug exposure
  * For 2 subjects who received the alternate treatment from which they were randomized, are switched to be analyzed according to actual treatment received
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 13 | 6
percentage of participants
  By 15 days (D16) | 46.15 | 83.33
  By 28 days (D29) | 76.92 | 100.00

17. Post Hoc Outcome: Time to Sustained Recovery Through Day 29 for Participant Sub-group With Interleukin-6 (IL-6) in the Highest Quartile (4th Quartile) at Baseline
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: Pooled Placebo vs Brilacidin 5-dose arm analyzed, for Post-hoc Per Protocol (PP) IL-6 sub-group.
  Post-hoc PP population is a subset of ITT population with the following differences:
  * Excludes subjects with viral load <10 copies/mL (i.e., below lower limit of quantitation) at baseline
  * Excludes subjects with <3 days of study drug exposure
  * For 2 subjects who received the alternate treatment from which they were randomized, are switched to be analyzed according to actual treatment received
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 12 | 9
percentage of participants
  By 15 days (D16) | 41.67 | 66.67
  By 28 days (D29) | 66.67 | 88.89

18. Post Hoc Outcome: Time to Sustained Recovery Through Day 29 for Participant Sub-group With SARS-CoV-2 Viral Load in the Highest Quartile (4th Quartile) at Baseline
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: Pooled Placebo vs Brilacidin 5-dose arm analyzed, for Post-hoc Per Protocol (PP) SARS-CoV-2 viral load sub-group.
  Post-hoc PP pop is a subset of ITT with the following differences:
  * Excludes subjects with viral load <10 copies/mL (i.e., below lower limit of quantitation) at baseline
  * Excludes subjects with <3 days of study drug exposure
  * For 2 subjects who received the alternate treatment from which they were randomized, are switched to be analyzed according to actual treatment received
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 11 | 13
percentage of participants
  By 15 days (D16) | 54.55 | 76.92
  By 28 days (D29) | 81.82 | 92.31

19. Post Hoc Outcome: Time to Sustained Recovery Through Day 29 for Participant Sub-group With Start of Study Treatment Within Fewer Than 7 Days of Onset of COVID-19 Symptoms
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: Pooled Placebo vs Brilacidin 5-dose arm analysis shown, for the Post-hoc Per Protocol (PP) sub-group starting study treatment <7 days from onset of COVID-19 symptoms.
  Post-hoc PP pop is a subset of ITT with the following differences:
  * Excludes subjects with viral load <10 copies/mL at baseline
  * Excludes subjects with <3 days of study drug exposure
  * For 2 subjects who received the alternate treatment from which they were randomized, are switched to be analyzed according to actual treatment
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo + SoC | Brilacidin 5-dose + SoC
Number analyzed (Participants) | 14 | 5
percentage of participants
  By 10 days (D11) | 35.71 | 60.00
  By 15 days (D16) | 50.00 | 100.00

ADVERSE EVENTS:
Time Frame: Day 1 through Day 60
Description: Adverse events are summarized for the safety population, which includes all subjects in the ITT population analyzed according to treatment received.
  Subjects treated with placebo were pooled for analyses since duration of placebo should not impact outcomes. As the different treatment durations for Brilacidin have potential to impact outcomes, 3-dose and 5-dose active arms were analyzed separately.
Groups:
- Total: Overall total
Arm/Group | Pooled Placebo + SoC | Brilacidin 3-dose + SoC | Brilacidin 5-dose + SoC | Total
All-Cause Mortality (participants affected / at risk) | 4/60 | 2/16 | 2/44 | 8/120
Serious Adverse Events (participants affected / at risk) | 7/60 | 3/16 | 4/44 | 14/120
Other Adverse Events (participants affected / at risk) | 39/60 | 14/16 | 39/44 | 92/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo + SoC (N=60) | Brilacidin 3-dose + SoC (N=16) | Brilacidin 5-dose + SoC (N=44) | Total (N=120)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 2 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo + SoC (N=60) | Brilacidin 3-dose + SoC (N=16) | Brilacidin 5-dose + SoC (N=44) | Total (N=120)
Alanine aminotransferase increased (Investigations) | 11 | 3 | 11 | 25
Aspartate aminotransferase increased (Investigations) | 8 | 2 | 5 | 15
Gamma-glutamyltransferase increased (Investigations) | 8 | 1 | 4 | 13
Blood pressure increased (Investigations) | 5 | 4 | 3 | 12
Serum ferritin increased (Investigations) | 3 | 0 | 4 | 7
Fibrin D dimer increased (Investigations) | 4 | 0 | 2 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 16 | 18
Hypoaesthesia oral (Nervous system disorders) | 0 | 1 | 9 | 10
Paraesthesia (Nervous system disorders) | 0 | 4 | 6 | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the disclosure agreement with investigators may vary. However, an investigator/institution may publish results, with any single center publication to be deferred until after a publication of results covering all centers in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT04784897/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04784897/SAP_001.pdf